CLINICAL TRIAL: NCT00890526
Title: Intervention for Reduced Sound Tolerance
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alabama, Tuscaloosa (Other)
Collaborators: University of Maryland (Other); University of Memphis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: DC004678; 7R01DC004678-06 (NIH)
Record Dates: First submitted 2009-04-28; First posted 2009-04-30 (Estimated); Last update posted 2012-06-21 (Estimated); Status verified 2012-06

CONDITIONS: Hyperacusis
Keywords: Tinnitus Retraining Therapy (TRT)
MeSH Terms: conditions — Hyperacusis | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Full treatment = Counseling + sound therapy.
  Interventions: Other: Sound Therapy (Tinnitus Retraining Therapy); Other: Counseling (Tinnitus Retraining Therapy)
- 2 (Experimental): Counseling + placebo sound therapy.
  Interventions: Other: Counseling (Tinnitus Retraining Therapy); Other: Placebo Sound Therapy
- 3 (Experimental): No Counseling + Sound Therapy
  Interventions: Other: Sound Therapy (Tinnitus Retraining Therapy); Other: No Counseling
- 4 (Placebo Comparator): No counseling + Placebo sound therapy.
  Interventions: Other: No Counseling; Other: Placebo Sound Therapy

INTERVENTIONS:
Other: Sound Therapy (Tinnitus Retraining Therapy) — The conventional sound therapy will be achieved with commercially available noise generators. Our clinic uses General Hearing Instruments (OHI) model Tranquil devices as noise sources for TRT. These flexible devices offer an adjustable volume control, with a frequency response extending from ~500 to 8000 Hz. Matched devices will be fitted binaurally and adjusted to each individual ear to achieve audibility of the noise sources (assessed by slight threshold shifts. typically 10- 15 dB, across the audiometric frequency range above 500 Hz). The sound pressure level output and frequency response of each noise source will be measured and documented using both real ear and standard electroacoustic methodologies. Each subject will be carefully instructed as to care of the instruments and correct volume setting. The bilateral noise generators will be used chronically during the intervention period except during sleep.
  Arms: 1; 3
Other: Counseling (Tinnitus Retraining Therapy) — The directive counseling to be used will include an in-depth participatory discussion with the patient to review audiometric and functional test results, along with the anatomy and physiology of the auditory system. A minimum of two hours will be scheduled to impart this information to the patients so that they will have a clear understanding of the disorder based upon the most current scientific data. The counseling will be focused on educating the patient, neutralizing their negative emotional association with the hyperacusis, and discussing their treatment.
  Arms: 1; 2
Other: No Counseling — Patients who are enrolled in Arms 3 and 4 of this study will not be offered directive counseling, but will be fitted with either conventional or placebo noise generators for their sound therapy components. These patients will be told only that their treatment for hyperacusis uses sound therapy. Otherwise, in the instrument fitting appointment (either for the conventional instrument or the placebo device), these patients will receive the same instruction in the care and use of sound generators as those patients enrolled in Treatment Arms 1 and 2 of the clinical trial.
  Arms: 3; 4
Other: Placebo Sound Therapy — The placebo sound therapy will use factory-modified GHI Tranquil noise generators, which will appear identical to the conventional Tranquil devices. The placebo Tranquil devices will have a control sensor installed to detect insertion of the device in the ear canal. When the sensor detects the insertion of the placebo device into the ear canal it will trigger gradual decay of the sound output from the placebo device, The time constant of the decaying noise output will be sufficiently long to allow the clinician time to set the volume of each binaural set of devices and to instruct the patient in their use before any noticeable sound attenuation occurs.
  Arms: 2; 4

SUMMARY:
Hyperacusis is the intolerance to sound levels that normally are judged acceptably loud to others. The presence of hyperacusis (diagnosed or undiagnosed) can be an important reason why some persons reject amplified sound from hearing aids. Tinnitus Retraining Therapy (TRT), originally proposed for the treatment of persons with debilitating tinnitus, offers the significant secondary benefit of increased Loudness Discomfort Levels (LDLs), along with expansion of the dynamic range for loudness. TRT uses both counseling and sound therapy from daily exposure to soft sound from bilateral noise generator devices (NGs) and has been promoted as an intervention for hyperacusis. The hypothesis of this investigational study is that the counseling and sound therapy principles used in TRT can be applied successfully to treat hearing-impaired hearing-aid candidates with reduced sound tolerance who are otherwise should benefit from hearing aids.

DETAILED DESCRIPTION:
Hyperacusis is the intolerance to sound levels that normally are judged acceptably loud to others. The presence of hyperacusis (diagnosed or undiagnosed) can be an important reason why some persons reject amplified sound from hearing aids. Tinnitus Retraining Therapy (TRT), originally proposed for the treatment of persons with debilitating tinnitus, offers the significant secondary benefit of increased Loudness Discomfort Levels (LDLs), along with expansion of the dynamic range for loudness. TRT uses both counseling and sound therapy from daily exposure to soft sound from bilateral noise generator devices (NGs) and has been promoted as an intervention for hyperacusis. The hypothesis of this investigational study is that the counseling and sound therapy principles used in TRT can be applied successfully to treat hearing-impaired hearing-aid candidates with reduced sound tolerance who are otherwise should benefit from hearing aids.

The current study is being implemented as a randomized, double-blind, placebo-controlled trial to assess the efficacy of a TRT-based intervention for reduced sound tolerance in hearing-aid eligible persons with hyperacusis and/or restricted dynamic ranges. The trial design allows for the evaluation of the efficacy of partial treatments, including the effects of counseling separately from the effects of sound therapy. Forty hearing-impaired subjects (without primary tinnitus) are being assigned randomly to one of four treatment groups: 1) full treatment, both counseling and sound-therapy (n=10); 2) counseling with placebo sound therapy (n=10); 3) sound therapy without counseling (n=10); and 4) placebo sound therapy without counseling (n=10). Subjects are being evaluated at least monthly, typically for five months or more, on a variety of audiometric tests, including LDLs, the Contour Test for Loudness for tones and speech, word recognition measured at each session's comfortable and loud levels, and electrophysiological measures.

ELIGIBILITY:
Inclusion Criteria:

* One hundred adults, who have hearing losses and who have unsuccessfully used hearing aids because of tolerance problems (hyperacusis).
* All subjects must be committed to the use of amplification if and when the hyperacusis is resolved.
* Each patient will have demonstrable hyperacusis, but will be free from tinnitus, and must be willing to wear and usc binaural in-the-ear sound generators (or placebo generators) chronically as prescribed.

Exclusion Criteria:

* Evidence of conductive, mixed hearing loss, or CNS disease.
* Abnormal tone and/or acoustic reflex decay will also preclude subject participation because of the potential for these patients to adapt to the chronic sound therapy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2002-07; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
>=dB-10 change in loudness discomfort level. | 5 consecutive monthly appointments

SECONDARY OUTCOMES:
Change in the contour 7. | 5 consecutive monthly appointments

CONTACTS AND LOCATIONS:
Locations (1):
- Univ. of Maryland - Baltimore, Baltimore, Maryland, United States